CLINICAL TRIAL: NCT07018180
Title: Interventional Study Evaluating the Use of COVER PATCH CAPTEUR PROTECT Support Solutions in Patients Living With Diabetes: a Prospective, Randomized, Controlled, Multicenter Study
Brief Title: Interventional Clinical Trial Evaluating COVER PATCH CAPTEUR PROTECT Support Solutions for Continuous Glucose Monitoring Sensors in Patients With Diabetes
Acronym: ICP-COVERPATCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CAPTEUR PROTECT (Industry)
Collaborators: Icadom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A01872-45
Record Dates: First submitted 2025-05-22; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Diabetes
Keywords: Diabetes; Continuous glucose monitoring; Adhesive patch; Cover patch; Poorly controlled
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVER PATCH (Experimental): Participants use their usual continuous glucose monitoring (CGM) sensor with the COVER PATCH adhesive patch during the study.
  Interventions: Device: Use of COVER patchs for continuous glucose monitoring sensor
- Standard of care (No Intervention): Participants use their usual continuous glucose monitoring (CGM) sensor without the COVER PATCH adhesive patch during the study (standard of care)

INTERVENTIONS:
Device: Use of COVER patchs for continuous glucose monitoring sensor — The intervention consists of wearing a patch over the continuous glucose monitoring (CGM) sensor typically used by the participant.
  The COVER patch is compatible with a wide range of CGM devices on the market, including Freestyle 2 or 3, Dexcom G6/One or G7/One+, and Guardian Sensor 4 or Simplera.
  At each sensor change, the participant is required to apply a new COVER PATCH over the CGM sensor. This is done throughout the entire duration of their participation in the study, which lasts for 4 months.
  Arms: COVER PATCH

SUMMARY:
The aim of this clinical trial is to evaluate whether the COVER PATCH adhesive patch can improve the adhesion of continuous glucose monitors (CGMs).

CGMs provide continuous blood sugar readings throughout the day and night, providing valuable data to help individuals manage their diabetes more efficiently. Many people face difficulties in keeping their CGM sensor in place.

Factors such as sweat, physical activity, heat, skin creams, and swimming can cause the sensor to fall off prematurely, interrupting glucose monitoring and making it harder to maintain stable blood sugar levels.

It has been shown that wearing a CGM sensor for at least 70% of the time is linked to better blood sugar control, measured by lower glycated hemoglobin (HbA1c). HbA1c reflects the average blood sugar over the past 3 months. A lower HbA1c level is associated with better diabetes management.

Currently, CGM sensors are designed for one-time use and need to be replaced every 7 to 15 days. However, when sensors fall off prematurely, they need to be replaced more frequently, leading to higher costs for patients. This can exceed what is covered by insurance. Some patients use non-approved solutions, like extra adhesive tapes, to keep their sensors in place, but these methods may not be effective.

This clinical trial aims to answer the following questions:

* Does the adhesive patch help keep the CGM sensor in place for the full recommended duration?
* Does better sensor adhesion lead to improved blood sugar control and lower HbA1c?
* Does the patch help reduce the frequency of premature sensor replacements?

To take part in this study, participants must be at least 6 years old and have type 1 or type 2 diabetes. Participants continue using their usual CGM during the study and are randomly assigned to either use the adhesive patch (COVER PATCH) or not. Participants and/or their parents (depending on the participant's age) complete questionnaires at the start of the study, and again at the end of the study at 4 months. Throughout the 4-month period, they also use an electronic tool (ePRO) to record each CGM sensor change and the reason for replacement.

This study may help improve how well glucose sensors stay in place, reduce the need to change them too often, and make it easier to manage blood sugar. It also aims to fulfill a medical need that is currently not adequately covered.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the effectiveness of COVER PATCH CAPTEUR PROTECT solutions for glucose sensors, in terms of improving glycemic control in patients with poorly controlled diabetes and suboptimal sensor wear time, compared to management without the COVER PATCH.

This is an interventional, prospective, randomized, controlled, multicenter clinical trial comparing the HbA1c levels of patients using COVER PATCH CAPTEUR PROTECT solutions for glucose sensors versus standard care.

The use of COVER PATCH CAPTEUR PROTECT solutions could result in a 0.3 percentage point improvement in HbA1c in diabetic patients initially having an HbA1c ≥ 8% and a glycemic sensor wear time of < 70%.

The device under study is the COVER PATCH solution by CAPTEUR PROTECT. This patch is a Class I, non-sterile, single-use device. COVER patches are intended for use in association with continuous glucose monitoring devices for patients living with diabetes.

COVER patches are compatible with a wide range of continuous glucose monitoring (CGM) devices available on the market. Several versions of the patches are available depending on the type of sensor (Freestyle 2 or 3, Dexcom G6/One or G7/One+, Guardian Sensor 4 or Simplera).

In this study, participants use their regular continuous glucose monitor (CGM), either with or without the adhesive patch being evaluated. Upon enrollment, retrospective data from the past 4 months are collected for analysis.

At the start of the study, participants complete the following questionnaires:

* Diabetes Treatment Satisfaction Questionnaire - status version (DTSQs)
* Diabetes Distress Scale (DDS) The adult, adolescent, or parent version is be provided depending on the participant's age.

Throughout the study, participants use an electronic tool (ePRO) to record each sensor change and indicate the reason for the replacement. Participants can also report any adverse events and device deficiency.

After 4 months, a follow-up visit takes place. Data from the previous 4 months are collected for analysis. Participants complete the same questionnaires again, as well as additional ones:

* Diabetes Treatment Satisfaction Questionnaire - change version (DTSQc)
* Physical activity questionnaire
* Satisfaction questionnaire regarding cover patch use The adult, adolescent, or parent version is be provided depending on the participant's age.

The study duration per patient is 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 6 years old
* Diagnosed with type 1 or type 2 diabetes
* Currently using a continuous glucose monitoring (CGM) sensor
* CGM sensor usage time < 70% over the last 4 months
* HbA1c ≥ 8% (verified by blood test or capillary test, no older than one month at the time of enrollment)
* Patient (or legal representative) owns a smartphone and has internet access (for completing questionnaires)
* Patient is covered by a social security scheme
* Patient (or legal representative, if applicable) is capable of reading and understanding the study procedure, and is able to give informed consent for participation in the study protocol

Exclusion Criteria:

* Patient with serious and untreated skin issues in the areas where the device will be applied (e.g., psoriasis, herpetiform dermatitis, skin rash, staphylococcal infection, etc.)
* Patient currently participating or having participated in an interventional clinical study within the month prior to enrollment that may impact the study, as determined by the investigator
* Patient or their legal representative who is deprived of liberty, under guardianship, or under curatorship.
* Pregnant or breastfeeding women, or women of childbearing age without an effective method of contraception, or those who do not agree to continue using contraception throughout the study duration. (Pregnancy will be checked by a urine HCG test for any woman wishing to participate and of childbearing age (under 60 years old).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the evolution of blood HbA1c, expressed in percentage points between enrollment and 4 months, in patients living with diabetes, with or without the COVER PATCH CAPTEUR PROTECT solution | 4 months

SECONDARY OUTCOMES:
Comparison of the average sensor wear time over 4 months, reported in percentage points relative to the duration of use claimed by the sensor manufacturers | 4 months
Comparison of the average sensor wear time, in days, over 4 months | 4 months
Comparison of the percentage (%) of patients for whom the sensor wear duration reached the maximum duration claimed by the manufacturer during the 4-month study period. | 4 months
Comparison of sensors' number used over 4 months | 4 months
Comparison of number change events for sensors, categorized by reason for change (detachment, loss of connection, etc.) at 4 months | 4 months
Comparison of change in scores of the Diabetes Treatment Satisfaction Questionnaire status at baseline (DTSQs) and at 4 months (DTSQs and DTSQc) | 4 months
  Adolescents (aged 12 to 17) will complete the age-appropriate version, the DTSQ-Teen. Parents of children aged 11 or younger will complete the parent version of the DTSQ (Parent-DTSQ)
  The DTSQ status (DTSQs) items are scored on a scale from 6 to 0 and DTSQ change (DTSQc) items are on a scale from 3 to -3.
  Higher is the score, the more the participant is satisfied (for DTSQs and DTSQc).
  DTSQs : The score ranges from 0 to 48 DTSQ parent : The score ranges from 0 to 84 DTSQ teen : The score ranges from 0 to 72 DTSQc Teen : The score ranges from -36 to 36 DTSQc Parent : The score ranges from -36 to 36 DTSQc : The score ranges from -24 to 24
Comparison of change in scores of the Diabetes Distress Scale (DDS) or the Parent Diabetes Distress Scale (Parent-DDS) at baseline and at 4 months | 4 months
  The DDS items are scored on a scale from 1 to 6. The score ranges from 1 to 6 (total score divided by the number of items) Higher is the score, the more living with diabetes is a burden for participant.
  The Parent-DDS items are scored on a scale from 1 to 5. The score ranges from 1 to 5 (total score divided by the number of items) Higher is the score, the more caring a children with diabetes is difficult for parents.
Assessment of the COVER PATCH CAPTEUR PROTECT satisfaction questionnaire, completed at 4 months | 4 months
  Satisfaction's evaluation : only for the interventional group, at 4 months Global satisfaction item with a scale from 1 to 5 Higher is the score, the more satisfied is the participant
Comparison of the percentage (%) of time spent in closed-loop mode | 4 months
  Only for participants in closed-loop
Comparison of the estimated HbA1c level (%) (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of the percentage (or average duration) of data captured (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of the percentage of time spent in the glucose range < 54 mg/dL (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of the percentage of time spent in the glucose range 54-69 mg/dL (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of the percentage of time spent in the glucose range 181-250 mg/dL (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of the percentage of time spent in the glucose range > 250 mg/dL (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of the percentage of time spent in the target glucose range 70-140 mg/dL (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of the average glucose level (mg/dL) (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of the daily glycemic coefficient of variation (collected from CGM plateforms, between baseline and 4 months) | 4 months
Comparison of adverse events' number, serious adverse events, adverse effects related to support solutions, and unexpected serious adverse effects related to support solutions occurring during the follow-up period | 4 months

CONTACTS AND LOCATIONS:
Locations (7):
- France (6):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU Grenoble Alpes, Grenoble
  - AP-HM Hôpital La Timone - Enfants, Marseille
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU Toulouse - Hôpital de Rangueil, Toulouse
- CHU Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No